CLINICAL TRIAL: NCT03190460
Title: Influence of Cognitive Training on Fall Prevention in At Risk Older Adults
Brief Title: Evaluating Technology-Based Fall Prevention Interventions
Acronym: FaCT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Hilaire Thompson, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 50219; R21NR015541 (NIH)
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Falls (Accidents) in Old Age
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Cognitive Training
- Education (Other)
  Interventions: Other: Technology-based Education

INTERVENTIONS:
Other: Cognitive Training — Web-based cognitive training intervention targeting specific cognitive tasks. Subjects complete 3 training sessions per week with at least 24 hours in between sessions.
  Arms: Intervention
Other: Technology-based Education — Subjects complete 16 web-based educational modules on healthy aging content. Following each module, subjects complete a learning reflection.
  Arms: Education

SUMMARY:
Approximately one in three older adults fall annually and it is the primary cause of traumatic injury in older adults. While exercise and balance programs have been shown to be effective in reducing fall risk, maintaining behavior change is known to be difficult. Thus additional interventions need to be validated to add to our current armamentarium to reduce falls in older adults. Cognitive training (CT) involves exercises that target specific cognitive tasks, such as memory or processing speed. It has been speculated that routinely performing such tasks may increase functional ability. Recent work has pointed to an increased risk of falls in community-dwelling older adults who have alterations in specific cognitive tasks. Thus the purpose of the proposed study is to demonstrate the feasibility and to explore the effectiveness of a 16 week CT intervention to reduce risk and incidence of fall and improve outcomes up to 1 month post-intervention in a group of community dwelling older adults at risk for fall.

ELIGIBILITY:
Inclusion Criteria:

* 65-89 years old
* speak and read English
* live within 30 miles of the University of Washington
* a score of 4 or higher on the Memory Impairment Screen (MIS-T)
* regular access to a computer with internet capability (whether at home, friend/family, community center, public library, or other)
* a positive response to any of the following three fall related questions: i) Have you had two or more falls in the prior 12 months? ii) Are you responding to the advertisement because of a recent fall? iii) Do you have difficulty with walking or balance?
* <53 seconds on 90 second balance test or gait speed <1m/sec.

Exclusion Criteria:

* current participation in formal cognitive training program
* currently bedridden or wheelchair dependent

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilaire Thompson, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson HJ, McGough E, Demiris G. Falls and Cognitive Training 2 (FaCT2) study protocol: a randomised controlled trial exploring cognitive training to reduce risk of falls in at-risk older adults. Inj Prev. 2020 Aug;26(4):370-377. doi: 10.1136/injuryprev-2019-043332. Epub 2019 Aug 26. PMID 31451566
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Education
Started | 40 | 20
Completed | 3 | 2
Not Completed | 37 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Education | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.2 (7.1) | 75.9 (6.6) | 76.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 44
  Male | 12 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 39 | 19 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 38 | 14 | 52
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Falls
Description: Falls and Injurious Falls as per Fall Calendar
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: number of falls
Arm/Group | Intervention | Education
Number analyzed (Participants) | 40 | 20
number of falls | 0.6 (0.2) | 0.6 (0.3)

2. Secondary Outcome: Disability
Description: Gill Disability Scale
Time Frame: 8 weeks, 16 weeks, 20 weeks.
Reporting Status: Not Posted

3. Secondary Outcome: Cognitive Assessment
Description: CANTAB Battery (Simple response time, one touch stockings of Cambridge, Stop Signal Task, Spatial Working Memory, Verbal Recognition Memory, Rapid Visual Information Processing)
Time Frame: 8 weeks, 16 weeks, 20 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Gait Assessment
Description: Assessment of Gait Parameters using APDM sensor system
Time Frame: 8 weeks, 16 weeks, 20 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Balance Assessment
Description: Assessment of Balance using APDM sensor system
Time Frame: 8 weeks, 16 weeks, 20 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Intervention | Education
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 0/40 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT03190460/Prot_SAP_001.pdf
  • Informed Consent Form (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03190460/ICF_000.pdf